CLINICAL TRIAL: NCT03837327
Title: Clinical Validation of the InterVenn Ovarian CAncer Liquid Biopsy (VOCAL)
Brief Title: Clinical Validation of the InterVenn Ovarian CAncer Liquid Biopsy
Acronym: VOCAL
Status: Completed | Type: Observational
Sponsor: Venn Biosciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: OVACA-001
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-08

CONDITIONS: Adnexal Mass; Ovarian Cancer; Pelvic Mass
Keywords: InterVenn; Ovarian Cancer; Liquid Biopsy; Mass Spectrometry; Adnexal Mass/ Pelvic Mass; Venn Biosciences; VOCAL Study
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adnexal Mass: Women with an adnexal mass (pelvic mass) as confirmed by imaging

SUMMARY:
Venn Biosciences Corporation ("InterVenn") has developed a liquid biopsy that is capable of distinguishing benign from malignant masses in women presenting with adnexal (pelvic) masses, through a simple blood test. The underlying technology combines mass spectrometry and artificial intelligence/machine learning to analyze tumor-associated changes in circulating glycoproteins.

The purpose of this study is to prospectively collect de-identified biological samples and data from women with a known pelvic mass, in order to validate ovarian cancer specific glycoproteomic signatures in the blood based on histologically confirmed malignancy status of the mass.

DETAILED DESCRIPTION:
This is a prospective, international, multi-center, observational study with a goal of collecting de-identified samples and data from 1,200 women with a known pelvic mass. Participants will consent to baseline and follow-up data and biospecimen collections.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years or older
* Able to provide a written informed consent and who understand and agree to all study procedures required
* A newly diagnosed adnexal mass as confirmed by imaging (computed tomography, ultrasonography, or magnetic resonance imaging) prior to enrollment
* Planned diagnostic procedure or surgery by the subject's physician to remove adnexal masses within 90 days of imaging. (Note that diagnostic procedure typically includes biopsy (needle core or laparoscopic-directed), ascites cytology, pleural effusion cytology or FNA)

Exclusion Criteria:

* Had/Has a diagnosis of invasive malignancy (exception: non-melanoma skin cancers) in the previous 5 years.
* Currently receiving or ever received any of the following prior cancer therapies in the previous 5 years. This includes curative surgical resection, local or systemic chemotherapy, targeted therapy, immunotherapy including cancer vaccines, hormone therapy, and/or radiation therapy.
* Pregnancy
* Current febrile illness
* Acute exacerbation or flare of an inflammatory condition requiring escalation in therapy
* Recipient of organ transplant
* Poor health status or unfit to tolerate blood draw

In addition, this study will include a small subgroup of women with a newly diagnosed clinically benign adnexal mass(es) for whom surgery is not planned as determined by the treating physician. This subgroup will follow the same exclusion criteria as listed above.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Per eligibility, individuals must have a known adnexal mass (pelvic mass).
Study Population: Adult women who present with a known adnexal mass as described in the study inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 1025 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
To determine the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of the VOCAL test | 24-48 Months

SECONDARY OUTCOMES:
To evaluate the association of protein and glycoprotein (GP) biomarkers with histological subtypes, stage, treatments and disease free survival (DFS) among woman with ovarian cancer | 24-48 Months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hommes, MD, Study Chair — InterVenn Biosciences
Locations (26):
- United States (10):
  - University of Southern California, Los Angeles, California
  - Bay Area Gynecology Oncology, San Jose, California
  - Palo Alto Medical Foundation, Sunnyvale, California
  - Mayo Clinic, Jacksonville, Florida
  - University of South Florida USF Health, OB/Gyn, Tampa, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Dr. Sudarshan K. Sharma, Ltd. - Gynecologic Oncology, Hinsdale, Illinois
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Optimum Clinical Research Group - Southwest Women's Oncology & Health, Albuquerque, New Mexico
  - Houston Methodist, Houston, Texas
- Royal Women's Hospital, Parkville, Victoria, Australia
- Malaysia (12):
  - Hospital Sultan Ismail, Johor Bahru, Johor
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Ampang, Ampang, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Taiping, Taiping, Perak
  - Hospital Seberang Jaya, Seberang Jaya, Pulau Pinang
  - Hospital Wanita Dan Kanak-kanak Sabah, Kota Kinabalu, Sabah
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Hospital Miri, Miri, Sarawak
  - Hospital Sibu, Sibu, Sarawak
  - Hospital Selayang, Batu Caves, Selangor
- Philippines (3):
  - The Medical City, Pasig, National Capital Region
  - National Kidney and Transplant Institute, Quezon City, National Capital Region
  - Philippine General Hospital, Manila